CLINICAL TRIAL: NCT04667351
Title: Hepatic Artery Infusion of Oxaliplatin, Leucovorin, and 2400 mg/m² Fluorouracil Versus Hepatic Artery Infusion of Oxaliplatin, Leucovorin, and 1200 mg/m² Fluorouracil for Unresectable Hepatocellular Carcinoma: a Randomised Phase 3 Non-inferiority Trial
Brief Title: HAIC of Oxaliplatin, and 2400 mg/m² 5-fu vs HAIC of Oxaliplatin, and 1200 mg/m² 5-fu for Unresectable HCC: a Randomised Phase 3 Non-inferiority Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Kaiping Central Hospital (Other); Guangzhou No.12 People's Hospital (Other Government)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SH-1
Record Dates: First submitted 2020-12-09; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: HepatoCellular Carcinoma
Keywords: Hepatic arterial infusion chemotherapy; 2400 mg/m² 5-fu; 1200 mg/m² 5-fu
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-fu 2400 (Active Comparator)
  Interventions: Drug: 2400 mg/m² 5-fu
- 5-fu 1200 (Experimental)
  Interventions: Drug: 1200 mg/m² 5-fu

INTERVENTIONS:
Drug: 2400 mg/m² 5-fu — Hepatic arterial infusion of oxaliplatin,leucovorin and 2400 mg/m² 5-FU
  Arms: 5-fu 2400
Drug: 1200 mg/m² 5-fu — Hepatic arterial infusion of oxaliplatin,leucovorin and 1200 mg/m² 5-FU
  Arms: 5-fu 1200

SUMMARY:
Hepatic artery infusion of oxaliplatin, leucovorin and 2400 mg/m² fluorouracil is effective in hepatocellular carcinoma. However, SILIUS study showed that sorafenib plus hepatic artery infusion of cisplatin and fluorouracil did not significantly improve overall survival compared with sorafenib alone. Whether fluorouracil is effevtive is known.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18-75 years;
* KPS≥70;
* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL).
* Patients must have at least one tumor lesion that can be accurately measured;
* Diagnosed as unresectable with consensus by the panel of liver surgery experts;
* No past history of TACE, HAIC, chemotherapy or molecule-targeted treatment;
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Meet the following laboratory parameters:(a) Platelet count ≥ 75,000/μL; (b)Hemoglobin ≥ 8.5 g/dL;(c) Total bilirubin ≤ 30mmol/L;(d) Serum albumin

  ≥ 32 g/L;(e) ASL and AST ≤ 6 x upper limit of normal;(f) Serum creatinine

  ≤ 1.5 x upper limit of normal;(g) INR > 2.3 or PT/APTT within normal limits; (h) Absolute neutrophil count (ANC) >1,500/mm3;
* Ability to understand the protocol and to agree to and sign a written informed consent document.

Exclusion Criteria:

* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known of serious heart disease which can nor endure the treatment such as cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Evidence of bleeding diathesis.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 24 months

SECONDARY OUTCOMES:
progression-free survival | 24 months
objective response rate | 6 months
disease control rate | 6 months
Adverse Events | 30 Days after HAIC

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Twelfth People 's Hospita, Guangzhou, Guangdong
  - Kaiping Central Hospital, Kaiping, Guangdong